CLINICAL TRIAL: NCT06791668
Title: Comparison of Different Regimens of Magnesium Sulphate in Patients With Severe Preeclampsia in Ain Shams University Maternity Hospital (Retrospective Cohort)
Brief Title: Different Regimens of Magnesium Sulphate in Patients With Severe Preeclampsia
Status: Recruiting | Type: Observational
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Rania Hassan Mostafa, Dr, Ain Shams University
Other Study IDs: FMASU MS 619/2024
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Preeclampsia (PE)
Keywords: eclampsia; magnesium sulphate; intensive care unit; pulmonary edema
MeSH Terms: conditions — Pre-Eclampsia; Eclampsia; Pulmonary Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- pregnant women with severe preeclampsia: Preeclampsia with severe hypertension that does not respond to treatment or is associated with ongoing or recurring severe headaches, visual scotomata, nausea or vomiting, epigastric pain, oliguria, and severe hypertension, as well as progressive deterioration in laboratory blood tests such as rising creatinine or liver transaminases or falling platelet count, or failure of fetal growth or abnormal doppler findings.

SUMMARY:
The goal of this observational study is to learn about the effects of the different drug regimens of magnesium sulphate in treatment of (severe pre-eclampsia). This condition affects some pregnant women and raises their blood pressure. It may also cause seizures (fits). The medication (magnesium sulphate) helps to prevent seizures. The main question this study aims to answer is:

What are the different regimens of magnesium sulphate that are used to prevent seizures in pregnant women with severe pre-eclampsia?

Participants already have taken the magnesium sulphate as part of their regular medical care for severe pre-eclampsia. Researchers will look into the records of the participants in the past 5 years to collect the data.

DETAILED DESCRIPTION:
This will be a retrospective study describing the different regimens of MgSO4 used in patients diagnosed with SPE in Ain Shams University Maternity Hospital (ASUMH), and the occurrence of eclamptic fits and any other complications with each of them.

Methodology:

1. Protocol approval will be sought from ethical committee and hospital administration.
2. Screening of all hospital records over the past 5 years to identify eligible records.
3. Eligible records will be reviewed to extract the following data:

   Age, Parity, Gestational age, BMI, Prior medical disorders, previous surgeries - including cesarean section (CS).

   Data upon admission: (Blood pressure, albuminuria) Available labs (CBC, AST, ALT, serum creatinine, PTT, INR) Timing (since admission) and route of delivery. Regimen of MgSO4 used (loading and maintenance doses, the route, and total time of therapy - antepartum and postpartum); any changes in dosage, and the reason for change.

   Any DOCUMENTED patient-reported MgSO4 side effects (nausea, vomiting, muscle weakness, palpitations, hypotension dizziness).

   Any DOCUMENTED signs of magnesium toxicity (clinical: defined as a presence of respiratory depression with less than 16 respirations per minute or loss of deep tendon reflexes necessitating cessation of MgSO4 or administration of calcium gluconate and / or biochemical: serum magnesium level >8.4mg/dl) Occurrence of eclamptic fits despite MgSO4 therapy, and timing, duration, how it was managed.

   Maternal admission to intensive care unit (ICU). Other complications (pulmonary edema, postpartum hemorrhage) Neonatal ICU (NICU) admission.

   All files with SPE will be examined. The number of files excluded from analysis will be noted as well as a table for the different causes of exclusion .

   Files showing serum magnesium level will be also analyzed in more detailed tables together with the reasons behind checking the serum level.
4. Data will be recorded in a case report form (appendix 1)
5. Statistical analysis will be done accordingly.

Ethical Consideration:

* The study design will be approved by the Local Ethics committee, Faculty of Medicine, Ain Shams University.
* Confidentiality will be respected in all levels of the study.

ELIGIBILITY:
Inclusion Criteria:

* All hospital records of patients diagnosed as preeclampsia with severe features planned to receive magnesium sulphate.

Exclusion Criteria:

* Records with missing data about the regimen of magnesium sulphate used

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital records will be reviewed for pregnant women presented to Ain Shams University Maternity Hospital (ASUMH) diagnosed as a case of preeclampsia with criteria of severity:
  Preeclampsia with severe hypertension that does not respond to treatment or is associated with ongoing or recurring severe headaches, visual scotomata, nausea or vomiting, epigastric pain, oliguria, and severe hypertension, as well as progressive deterioration in laboratory blood tests such as rising creatinine or liver transaminases or falling platelet count, or failure of fetal growth or abnormal doppler findings.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Occurrence of eclamptic fits | within 24 hours before or after delivery
  Development of generalized tonic clonic convulsions in pregnant women with preeclampsia

SECONDARY OUTCOMES:
ICU admission | within 48 hours before or after delivery
  admission to the intensive care unit
magnesium sulphate toxicity | within 48 hours before or after delivery
  clinical: defined as a presence of respiratory depression with less than 16 respirations per minute or loss of deep tendon reflexes necessitating cessation of MgSO4 or administration of calcium gluconate and / or biochemical: serum magnesium level >8.4mg/dl
primary postpartum hemorrhage | within 24 hours after delivery
  occurrence of complications as primary postpartum hemorrhage (the loss of 500 ml or more of blood from the genital tract within 24 hours of the birth of a baby)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the dataset generated and analyzed in this study after publication of the results.
Supporting Information: Study Protocol, Analytic Code
Time Frame: start date: after publication of the study results end date: for 10years